CLINICAL TRIAL: NCT04659486
Title: Prospective Studies in School-aged Children and Adolescents With COVID-19 Treated at HCFMUSP
Brief Title: Adolescents With COVID-19/MIS-C at HCFMUSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Sao Paulo (Other)
Collaborators: Hospital das Clínicas da Faculdade de Medicina da USP (Unknown); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 37460620.8.0000.0068
Record Dates: First submitted 2020-12-01; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Covid19; Corona Virus Infection; SARS (Severe Acute Respiratory Syndrome); SARS-CoV Infection
Keywords: Covid19; Children; Adolescents
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training (Experimental): A 12 weeks parallel-group randomized controlled trial will be performed, in which covid-19 survivors adolescents will complete a telemonitored home-based exercise training program, 3 times per week. The training program will involve strength and aerobic exercises
  Interventions: Behavioral: Home-based exercise training
- Control (No Intervention): The control group will receive all regular medical care and advice on healthy lifestyle including the promotion of recommended physical activity levels.

INTERVENTIONS:
Behavioral: Home-based exercise training — Online strength and aerobic home-based exercise training, 3 times per week, for 12 weeks. The exercise program is composed by 2 intensity-levels (starter and advanced).
  Arms: Exercise training

SUMMARY:
This is a protocol aimed at children and adolescents contaminated with COVID, treated at the Hospital das Clínicas, University of Sao Paulo, Brazil (HCFMUSP), in the recovery phase. The study aims to evaluate the spectrum of pathogenic lesions of the virus not only in the respiratory system, but digestive, immunological, neurological and others. Clinical, evolutionary, laboratory and functional parameters will be used.

DETAILED DESCRIPTION:
School-age children and adolescents COVID-19 survivors may have persistent inflammation, a chronic course of COVID-19, with isolated or concomitant aggressions of various organs and systems, making this disease a potential chronic condition, impacting aspects of quality of life related to health (HRQoL), physical and mental health. In addition, pediatric COVID-19 can induce autoimmunity (with the possibility of primary hypothyroidism and type I diabetes mellitus), delayed linear growth and delayed pubertal development, secondary immunodeficiency and present genetic polymorphisms in brain plasticity impacting rehabilitation. School-aged children and adolescents with COVID-19 could present muscle weakness, dysautonomy, asthenia and physical inactivity, so it is essential that safe and effective interventions are developed to maintain adequate levels of physical activity and that they can be implemented on a large scale. However, to date, there are no systematic longitudinal studies that have evaluated all these aspects in a pediatric population that survived COVID-19, particularly with chronic conditions and who were hospitalized in a tertiary service.

ELIGIBILITY:
Inclusion Criteria:

* school-age children and adolescents diagnosed with COVID-19

Exclusion Criteria:

* school-age children and adolescents with MIS-C, who present: myocardial dysfunction, refractory cardiac arrhythmias, coronary artery aneurysms with or without thrombi, electrocardiographic alterations suggestive of myocardial infarction or ischemia and clinical signs of heart failure;
* presence of any limitation or physical disability that prevents the practice of exercise;
* pregnancy.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life assessed by the Pediatric Quality of Life Inventory (Peds-QoL) | Change from Baseline at 3 months
  The instrument was translated and validated for the Brazilian population
Quality of Life assessed by the Pediatric Quality of Life Inventory (Peds-QoL) | Change from Baseline at 6 months
  The instrument was translated and validated for the Brazilian population

SECONDARY OUTCOMES:
Flow-volume loop assessed by spirometry | Baseline, 3 months, 6 months
  Aims to investigate the mechanisms that lead to dyspnea and, consequently, intolerance to physical effort
Health-related quality of life assessed by the Pediatric Outcomes Data Collection Instrument | Baseline, 3 months, 6 months, 12 months
  It will also be assessed for school-age children (7-10 years old) and adolescents (11-18 years old) and by their primary caregiver
Complete blood count (hemoglobin, leukocyte, lymphocyte and platelet count) | Baseline, 3 months, 6 months, 12 months
Inflammatory markers (C-reactive protein, fibrinogen, D-dimer and ferritin); | Baseline, 3 months, 6 months,12 months
Lactate dehydrogenase | Baseline, 3 months, 6 months, 12 months
Aspartate and alanine aminotransferase | Baseline, 3 months, 6 months, 12 months
Serum urea and creatinine | Baseline, 3 months, 6 months, 12 months
Triglycerides | Baseline, 3 months, 6 months, 12 months
Creatinine phosphokinase (CK) | Baseline, 3 months, 6 months, 12 months
Amilase | Baseline, 3 months, 6 months, 12 months
Lipase | Baseline, 3 months, 6 months, 12 months
Troponin T | Baseline, 3 months, 6 months, 12 months
Pro-BNP | Baseline, 3 months, 6 months, 12 months
Lung abnormalities will be assessed by pulmonary computed tomography | Baseline, 3 months, 6 months, 12 months
  Patchy ground-glass opacities, crazy-paving pattern, and localization and pattern of large, confluent or small nodular lesions will be assessed
Systolic and diastolic function will be assessed by echocardiogram | Baseline, 3 months, 6 months, 12 months
  Conventional transthoracic echocardiogram with color Doppler to assess systolic and diastolic function
Valve dysfunction will be assessed by echocardiogram | Baseline, 3 months, 6 months, 12 months
  Conventional transthoracic echocardiogram with color Doppler to search for valve dysfunction
Pericardial effusion will be assessed by echocardiogram | Baseline, 3 months, 6 months, 12 months
  Conventional transthoracic echocardiogram with color Doppler to search for pericardial effusion
Coronary arteries will be assessed by echocardiogram | Baseline, 3 months, 6 months, 12 months
  Conventional transthoracic echocardiogram with color Doppler to search for aspects of the coronary arteries
Ischemia will be assessed by echocardiogram | Baseline, 3 months, 6 months, 12 months
  Echocardiogram with two-dimensional speckle-tracking technique to identify subclinical changes suggestive of ischemia or myocarditis
Immunocompetence, including thymic function | Baseline, 3 months, 6 months, 12 months
  Baseline levels of cytokines IL-2, IL-4, IL-6, IL-10, TNF-alpha, IFN-y, and IL-17A in serum samples will be tested by flow cytometry using the CBA technique (Cytometric bead array, BD Biosciences)
Leukogram will be assessed by leukocyte and lymphocyte counts | Baseline, 3 months, 6 months,, 12 months
Immunophenotyping of lymphocytes T cell lineages will be evaluated by flow cytometry | Baseline, 3 months, 6 months, 12 months
  T cell lineages: CD3CD4, CD3CD8, naive cells (CD45RA+), memory cells (CD45RA-), effector cells (CD38+HLADR+)
Immunophenotyping of lymphocytes B cell lineages will be evaluated by flow cytometry | Baseline, 3 months, 6 months, 12 months
  B cell lineages: CD19, naive cells (CD27-), memory cells (CD27+), plasmablasts (CD27+CD38+CD138-), (plasmocytes CD27+CD38+CD138+)
Immunophenotyping of lymphocytes NK cells will be evaluated by flow cytometry | Baseline, 3 months, 6 months, 12 months
  NK cells: (CD3-CD16+CD56+), degranulated: CD107a+
Serum levels of anti-Streptococcus pneumoniae IgG antibodies | Baseline, 3 months, 6 months, 12 months
Anti-pneumococcal vaccine response will be assessed by ELISA | Baseline, 3 months, 6 months, 12 months
  The antipneumococcal antibody titer against 6 polysaccharides (serotypes 1, 5, 6B, 9V, 14, and 18C) will be analyzed by ELISA. The seroconversion criteria is IgG values > 1.3 mg/mL for each polysaccharide assessed
Evaluation of the thymus by the determination of TRECs (Thymic recent emigrant cells or T-cell receptor excision circles) | Baseline, 3 months, 6 months, 12 months
  TRECs evaluate the peripheral function of the thymus from cells that have recently been released, using the RT-PCR technique
Changes in frequency of the autoantibodies of the thyroid gland | Baseline, 3 months, 6 months, 12 months
  (anti-thyroperoxidase antibodies, anti-thyroglobulin)
Changes in frequency of the anti-GAD antibody will be assessed using immunoprecipitation | Baseline, 3 months, 6 months, 12 months
Changes in frequency of the anti-islet antibody of Langerhans will be assessed using indirect fluorescence | Baseline, 3 months, 6 months, 12 months
Changes in frequency of the anti-insulin antibody will be assessed by radioimmunoassay | Baseline, 3 months, 6 months, 12 months
Diagnosis of thyroid dysfunction will be assessed by thyroid profile (TSH, free T4 and T3) | Baseline, 3 months, 6 months, 12 months
Diagnosis of type 1 diabetes mellitus will be assessed by the metabolic profile (fasting glucose, glycated hemoglobin and C peptide) | Baseline, 3 months, 6 months,, 12 months
Linear growth will be assessed by using a standardized stadiometer, calculating standard deviation, growth curves, and growth speed | Baseline, 3 months, 6 months, 12 months
Development of puberty will be assessed according to the criteria of Tanner and Marshall in adolescents in the prepubertal age group | Baseline, 3 months, 6 months, 12 months
Bone age will be assessed using non-dominant hand and wrist radiography | Baseline, 12 months
Bone mineral density will be assessed by Bone densitometry (DXA) in the region of the lumbar spine | Baseline, 3 months, 6 months, 12 months
Bone mineral content will be assessed by Bone densitometry (DXA) in the region of the lumbar spine | Baseline, 3 months, 6 months, 12 months
Bone mineral density will be assessed by Bone densitometry (DXA) in the proximal femur | Baseline, 3 months, 6 months, 12 months
Bone mineral content will be assessed by Bone densitometry (DXA) in the proximal femur | Baseline, 3 months, 6 months, 12 months
Bone mineral density will be assessed by Bone densitometry (DXA) in the whole body | Baseline, 3 months, 6 months, 12 months
Bone mineral content will be assessed by Bone densitometry (DXA) in the whole body | Baseline, 3 months, 6 months, 12 months
Body composition (visceral adipose tissue) will be assessed by Bone densitometry | Baseline, 3 months, 6 months, 12 months
Body composition (lean mass) will be assessed by Bone densitometry | Baseline, 3 months, 6 months, 12 months
Body composition (fat mass) will be assessed by Bone densitometry | Baseline, 3 months, 6 months, 12 months
Bone biochemical and bone remodeling markers (calcium, phosphorus, 25OH alkaline phosphatase vitamin D, PTH, CTX, P1NP) | Baseline, 3 months, 6 months, 12 months
Pediatric gait assessment will be assessed by an Actigraph (3D accelerometer) model G-Walk used during the "timed up and go" test | Baseline, 3 months, 6 months, 12 months
Pediatric gait assessment will be assessed by an Actigraph (3D accelerometer) model G-Walk during the 6-minute walk test | Baseline, 3 months, 6 months, 12 months
Pediatric gait assessment will be assessed by an Actigraph (3D accelerometer) model G-Walk during the 10 meter gait test | Baseline, 3 months, 6 months, 12 months
Pediatric gait assessment will be assessed by musculoskeletal ultrasound | Baseline, 3 months, 6 months, 12 months
Genetic Polymorphism Analysis will be assessed by salting out methodology followed by q-PCR (Real-time PCR) using the TaqMan assay using Step One Plus equipment | Baseline, 3 months, 6 months, 12 months
  According to the gene sequence studied, the analysis will be performed using the Sanger sequencing technique with capillary electrophoresis in a 3130 automatic sequencer (Applied Biosystems).
  The genetic polymorphisms of the ABO system gene (rs505922), two polymorphisms of the OPRM1 gene (rs1799971 and rs1799972) and a polymorphism of the BDNF gene (rs6265) will be investigated, with possible contributions to the risk of impaired gait.
Mental health will be assessed by the "Strengths and Weaknesses of Attention-deficit/hyperactivity disorder (ADHD) symptoms and Normal behaviors" | Baseline, 3 months, 6 months, 12 months
  This is an 18-item parent questionnaire for children and adolescents (18 years and younger). This rating scale includes positive "weaknesses" and negative "strengths" scoring, assessing symptoms of Attention-Deficit/Hyperactivity Disorder. Parents are asked to compare their child's behavior in a variety of settings over the past month to other children on a 7-point: 3-Far below, 2-Below, 1-Slightly below, 0-Average, -1-Slightly average, -2-Above, -3-Far above. Higher scores indicate greater symptomology
Mental health will be assessed by the "Strengths and Difficulties Questionnaire" | Baseline, 3 months, 6 months, 12 months
  The Strengths and Difficulties Questionnaire (SDQ) is a brief behavioural screening questionnaire, and includes 25 items on psychological attribute: emotional symptoms (5 items), conduct problems (5 items) hyperactivity/inattention (5 items), peer relationship problems (5 items), prosocial behaviour (5 items). Higher scores indicate greater difficulties
Mental health will be assessed by the "Depression, Anxiety and Stress Scale" | Baseline, 3 months, 6 months, 12 months
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress (7 items each subscale). Patients are asked to score every item on a scale from 0 (did not apply to me at all) to 3 (applied to me very much). Sum scores for the total DASS-total scale range between 0 and 120. Scores ≥60 (for DASS-total) and ≥21 (for the depression subscale) are labeled as "high" or "severe".
Physical activity levels assessed by ActivPAL | Baseline, 3 months, 6 months, 12 months
  ActivPAL will be used for 7 days for at least 10 hours/day
Food consumption levels assessed by food records | Baseline, 3 months, 6 months, 12 months
  24-hour recalls will be assessed on three non-consecutive days (two weekdays, and one weekend). Online Dietbox will be used.
Blood flow will be assessed using a Doppler Ultrasound | Baseline, 3 months, 6 months, 12 months
  Baseline blood flow measurements will be assessed in the brachial artery
Endothelial function will be assessed using a Doppler Ultrasound | Baseline, 3 months, 6 months, 12 months
  Flow-mediated vasodilation (VMF) will be assessed in the brachial artery

CONTACTS AND LOCATIONS:
Overall Officials: Clovis Silva, PhD, Study Director — University of Sao Paulo
Locations (1):
- Hospital das Clinicas Faculdade de Medicina USP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Astley C, Drezner JA, Sieczkowska SM, Ihara A, Franco T, Gil S, DO Prado DML, Longobardi I, Suguita P, Fink T, Lindoso L, Matsuo O, Martins F, Bain V, Leal GN, Badue MF, Marques HH, Silva CA, Roschel H, Gualano B. Exercise in Pediatric COVID-19: A Randomized Controlled Trial. Med Sci Sports Exerc. 2025 Mar 1;57(3):514-523. doi: 10.1249/MSS.0000000000003589. Epub 2024 Nov 6. PMID 39501479